CLINICAL TRIAL: NCT04963673
Title: Evaluation of Interaction Between Immunosuppressive Drugs and Protein-bound Uremic Toxins in Renal Transplant Patients
Acronym: DRUGTOX
Status: Withdrawn | Type: Observational
Why Stopped: no participants enrolled
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2019_843_0060
Record Dates: First submitted 2021-07-06; First posted 2021-07-15 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Kidney Transplant; Immunosuppression; Uremic; Toxemia
Keywords: Kidney Transplant; Immunosuppression; Uremic; Toxemia
MeSH Terms: conditions — Toxemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DFG> 40 ml / min: Kidney transplant population followed at CHU Amiens (group 1 ⇾ DFG> 40 ml / min).
  Interventions: Other: calcineurin inhibitor dosage
- DFG < 40 ml / min: Kidney transplant population followed at CHU Amiens (group 2 ⇾ DFG < 40 ml / min).
  Interventions: Other: calcineurin inhibitor dosage

INTERVENTIONS:
Other: calcineurin inhibitor dosage — The dosage of calcineurin inhibitors will be done as usual by the toxicology pharmacology laboratory of the CHU Amiens-Picardie. If the patient does not object, the determination of protein-bound uremic toxins from the rest of the collected blood tube will be performed using high performance liquid chromatography.

SUMMARY:
The majority of studies conducted on uremic toxins involve patients before end stage renal failure or dialysis patients. Only a few studies have focused on transplant patients. In addition, the relationship between serum concentrations of uremic toxins and immunosuppressive drug concentrations has never been studied to date.

The investigator research hypothesis is that, due to the strong plasma protein binding of calcineurin inhibitors, an interaction with protein-bound uremic toxins could alter drug concentrations that explain difficulties in reaching therapeutic targets.

DETAILED DESCRIPTION:
In France, the national prevalence of end-stage kidney disease (including dialysis and renal transplantation) is 1,232 per million inhabitants. As in all transplants, renal transplantation needs immunosuppressive therapy. This treatment may be difficult to adjust in some patients. However, achieving the therapeutic target is essential to have an efficiency synonymous with graft survival and better tolerance to the drug. The immunosuppressive class drug of interest in the present project is the class of calcineurin inhibitors (tacrolimus and ciclosporin) that are widely used in both initial and maintenance immunosuppression. These drugs have the pharmacological specificities to be highly bound to plasma proteins and requiring pharmacological therapeutic monitoring.

With the progression of chronic kidney disease, many molecules accumulate as a result of decreased kidney excretion capacity, such as compounds called uremic toxins. The investigators research is part of the European network for the study of these toxins (Eutox group) and has largely contributed to the better knowledge of these toxins. In particular, they are defined by their dose-dependent deleterious effects. These molecules are classified, according to their molecular weight, into small molecules, medium molecules and molecules strongly bound to plasma proteins (p-cresyl sulphate [pCS], indoxyl sulphate [IS] and indol acetic acid [IAA]). This last group of protein will be evaluated in this project.

The majority of studies conducted on uremic toxins involve patients before end stage renal failure or dialysis patients. Only a few studies have focused on transplant patients. In addition, the relationship between serum concentrations of uremic toxins and immunosuppressive drug concentrations has never been studied to date.

the investigator research hypothesis is that, due to the strong plasma protein binding of calcineurin inhibitors, an interaction with protein-bound uremic toxins could alter drug concentrations that explain difficulties in reaching therapeutic targets.

ELIGIBILITY:
Inclusion Criteria:

* renal transplant patient followed at the University Hospital of Amiens and transplanted for over a year
* patient treated with a calcineurin inhibitor
* patient having a blood test for evaluation of calcineurin inhibitor concentrations by the toxicology pharmacology laboratory of the Amiens-Picardie University Hospital,
* patient affiliated with social security.

Exclusion Criteria:

* patient in phase of acute rejection of the graft,
* patient having opposed his participation,
* patient under guardianship or curatorship or deprived of public right

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney transplant population followed at CHU Amiens (group 1 ⇾ DFG> 40 ml / min, group 2 ⇾ DFG < 40 ml / min).
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-07-06 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
plasma tacrolimus concentration without plasma uremic toxin adjustment | at day 0
plasma tacrolimus concentration with plasma uremic toxin adjustment | at day 0

SECONDARY OUTCOMES:
plasma ciclosporin concentration without plasma uremic toxin adjustment | at day 0
plasma ciclosporin concentration with plasma uremic toxin adjustment | at day 0

CONTACTS AND LOCATIONS:
Overall Officials: Youssef Bennis, MD, Principal Investigator — CHU Amiens; Sandra Bodeau, MD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No